CLINICAL TRIAL: NCT06282198
Title: Evaluating Functional Outcomes and Quality of Life in Musculoskeletal Tumor Patients With Distal Femoral Megaprostheses: A Case-Control Study
Brief Title: Functional Outcomes and Quality of Life in Musculoskeletal Tumor Patients With Distal Femoral Megaprostheses
Acronym: FOQ-DFP
Status: Completed | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Chair Profesor, Cardenal Herrera University
Other Study IDs: UCHCEU-13/02/24
Record Dates: First submitted 2024-02-13; First posted 2024-02-28 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Distal Femoral Musculoskeletal Tumors
Keywords: Megaprosthesis; Musculoskeletal tumor; Distal femur; Lower limb; Functional mobility; Quality of life; Case-Control Study; Inertial Measurement Unit

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with Distal Femoral megaprosthesis
- Control: Healthy subjects

SUMMARY:
This study aims to evaluate the functional outcomes of patients with distal femur tumor prostheses in comparison to a matched control group.

DETAILED DESCRIPTION:
The aim of this case-control study will be to compare functional outcomes-including results from the TUG and 6MWT, knee flexor and extensor muscle strength, sagittal knee range of motion-and health-related quality of life between patients with distal femoral megaprostheses and healthy controls. By employing both traditional assessments and IMU technology, the investigators will provide a comprehensive evaluation of functional recovery in this population, thereby informing clinical practice and rehabilitation strategies.

Two functional tests that will be conducted are the Time Up and Go Test and the 6-Minute Walk Test. These tests will be administered using a non-invasive Inertial Measurement Unit (IMU), specifically the BTS G-sensor inertial sensor (BTS Bioengineering, Garbagnate Milanese, Italy), positioned at the S1 level to collect spatiotemporal gait data. These data will then be analyzed in comparison to values obtained from healthy participants.

The assessment will include anamnesis and a complete clinical examination of tumor patients with distal femur megaprostheses undergoing surgery at Hospital la Fe in Valencia, focusing on knee joint mobility and muscle group strength. Subjective function will be evaluated using questionnaires such as the SF-36 for both cases and controls and the MSTS (Musculoskeletal Tumor Society Score) for cases.

ELIGIBILITY:
Inclusion Criteria (cases group):

* Megaprosthesis of unilateral distal femur
* Tumor cause
* Ambulation capacity

Exclusion Criteria (cases group):

* Neurological alterations prior to the inervention than affect the lower limbs or general movement
* Patient incapable of ambulation due to progression of his/her pathology
* Patient with palliative treatment for advanced tumor diseas
* More than one ipsilateral or contralateral prosthesis
* Infection, traumatic or sequel to revision surgery cause

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cases: Patients with megaprosthesis of the distal femur due to tumor treated at Hospital Universitario la Fe.
  Controls: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
SF-36 questionnaire | 3 months
  This instrument assesses health-related quality of life and comprises 36 items, organized into eight subscales: physical functioning (10 items), physical role functioning (4 items), bodily pain (2 items), general health perceptions (5 items), vitality (4 items), social functioning (2 items), emotional role functioning (3 items), and mental health (5 items). Each subscale is scored on a scale from 0 to 100, with higher scores indicating better health status in that domain.
  In addition to individual subscale scores, two aggregate summary scores are calculated: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). These summary scores are norm-based, with a mean of 50 and a standard deviation of 10, allowing comparison to population averages. Scores above 50 represent better-than-average health, while scores below 50 indicate lower-than-average health-related quality of life.
Timed Up and Go Test | 3 months
  Participants are seated in a chair with their backs against the backrest and their hands resting on their thighs. Upon the verbal command "GO", they are instructed to stand, walk down a 3-meter pathway, turn around, and return to a seated position as quickly and safely as possible. The recorded parameters include total TUG time (s), rotation speed during the middle and final turns (°/s), and vertical acceleration during the sit-to-stand and stand-to-sit transitions (m/s²)
6 -Minute Walk Test | 3 months
  This test is conducted in a continuous 30-meter corridor, where participants are instructed to walk for 6 minutes at their own preferred pace. The primary parameter measured is total walking distance (m)

SECONDARY OUTCOMES:
Sagittal range of movement of the knee measured with a goniometer | 3 months
  Sagittal range of movement of pathologic knee and healthy knee in controls.Full knee extension is considered 0º. The full range of knee mobility determined by the sum of the degrees of flexion plus the degrees of extension.
Muscular strength | 3 months
  We measure muscle strength in the quadriceps and hamstrings of the pathological leg in the cases and one of the legs in the controls. For this we use the Medical Research Council Scale.
  On this scale, contraction is assessed from 0-5.
  Grade 5: Normal
  Grade 4: Movement against gravity and resistance
  Grade 3: Movement against gravity over (almost) the full range
  Grade 2: Movement of the limb but not against gravity
  Grade 1: Visible contraction without movement of the limb
  Grade 0: No visible contraction
MSTS Score | 3 months
  Musculoskeletal Tumour Society (MSTS) Score evaluates patients' subjective functional capabilities. This assessment comprises six subscales: pain, function, emotional acceptance, use of assistive devices for ambulation, walking ability, and gait. Each subscale is rated on a scale from 0 to 5 points, with 5 indicating the most favorable outcome. Total scores are categorized as follows: poor (<15%), fair (15-17%), moderate (18-20%), good (21-22%), and excellent (23-30%). Higher total scores reflect better functional performance

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Lisón, PhD, Study Director — Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided